CLINICAL TRIAL: NCT04030377
Title: Treatment of Postoperative Urinary Retention - WHAT DO WOMEN WANT?
Brief Title: Postop Catheterization for Urinary Retention
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment, question addressed by other researchers
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Other Study IDs: EH11-096
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates patient's preference and satisfaction with choice of catheterization after surgical urogynecological procedures.

DETAILED DESCRIPTION:
Preoperatively, the enrolled patient receives information about risks and benefits of three ways of bladder catheterization as means of management of postoperative urinary retention. Based on this information, the patient chooses her preferred way of postoperative catheterization in case she experiences acute urinary retention after surgery. After the surgery, those patients requiring catheterization postoperatively evaluate their experience in a postoperative questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All female patients who undergo urogynecological surgery procedures at NorthShore University HealthSystem and consent to participate

Exclusion Criteria:

* Patients who cannot read, comprehend, and write in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women presenting to the urogynecology offices at NorthShore University HealthSystem with a urogynecologic diagnosis desiring surgical management.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with choice of catheterization method | 2 weeks after index procedure
  Assessed through post-operative questionnaire completion

SECONDARY OUTCOMES:
Assessment of complication rates | 2 weeks after index procedure
  Comparison of complication rates between intermittent vs. indwelling catheterization: data derived from review of participant medical record

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia M Botros, MD, Study Director — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Skokie, Illinois, United States